CLINICAL TRIAL: NCT02596789
Title: Study of Cortical Excitability in Healthy Subjects With Transcranial Magnetic Stimulation (TMS) and a Neuronavigation Device
Brief Title: Cortical Excitability Using Transcranial Magnetic Stimulation and Neuronavigation Device
Acronym: RC-TMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-A00316-37
Record Dates: First submitted 2014-07-23; First posted 2015-11-04 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- state dependency TMS (Other): TMS performed at rest and during a cognitive/emotional task
  Interventions: Device: TMS "Magpro®, Magventure Inc" device

INTERVENTIONS:
Device: TMS "Magpro®, Magventure Inc" device

SUMMARY:
This study has two main goals :

* to investigate the impact of aging on cortical excitability (CE)
* to investigate the impact of "state dependency" on CE, using a cognitive task and an emotional one.

A Neuronavigation system of transcranial magnetic stimulation is used, and electromyographic response are recorded.

ELIGIBILITY:
Inclusion Criteria:

* male or female
* age 18-75
* signed informed consent
* normal physical examination

Exclusion Criteria:

* less 18 or more 75 years of age
* contra indication to TMS: epilepsia or seizures, metallic head devices, cardiac pacemaker, pregnancy, jet lag or severe insomnia the night before
* severe physical disease
* treatment with psychotropic drugs
* overt psychiatric disease
* alcohol consumption before the examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Amplitudes of Motor evoked Potentials (µV) for ICI and ICF. | Participants will be followed for an expected average of one month
  Motor Evoked Potential (MEP) from the first dorsal interosseous are register during the stimulations.
  Intracortical Inhibition (ICI) and Facilitation (ICF) are a paired-pulse TMS measure of cortical excitability. A short Interval interstimuli (2ms) leads to a cortical inhibition, which reflects the GABAergic neurotransmission; whereas a longer interval interstimuli leads to a cortical facilitation, which reflects glutamatergic neurotransmission.
Durations of Cortical Silent Period (ms) | Participants will be followed for an expected average of one month
  Cortical Silent Period (CSP) is a single-pulse TMS measure of cortical inhibition, stimulations are applied while subjects are exerting a muscular contraction of the thum-index pinch and lead to a muscular cancellation. Duration of this silence is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry BOUGEROL, MD, PhD, Principal Investigator — University of Grenoble
Locations (1):
- Department of Psychiatry & Neurology - University Hospital Grenoble, Grenoble, France